CLINICAL TRIAL: NCT02541565
Title: MK-3475 in Combination With Standard RCHOP Therapy for Previously Untreated Diffuse Large B-Cell Lymphoma
Brief Title: Pembrolizumab and Combination Chemotherapy in Treating Patients With Previously Untreated Diffuse Large B-cell Lymphoma or Grade 3b Follicular Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9291; NCI-2015-01309 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MK-3475; 9291 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-08

CONDITIONS: Composite Lymphoma; Grade 3b Follicular Lymphoma; Stage I Diffuse Large B-Cell Lymphoma; Stage I Follicular Lymphoma; Stage II Diffuse Large B-Cell Lymphoma; Stage II Follicular Lymphoma; Stage III Diffuse Large B-Cell Lymphoma; Stage III Follicular Lymphoma; Stage IV Diffuse Large B-Cell Lymphoma; Stage IV Follicular Lymphoma
MeSH Terms: conditions — Composite Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Cyclophosphamide; Doxorubicin; pembrolizumab; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, combination chemotherapy) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and prednisone PO on days 1-5. Patients also receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 2 of course 1 and on day 1 of subsequent courses. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This pilot phase I trial studies the side effects of pembrolizumab and combination chemotherapy in treating patients with previously untreated diffuse large B-cell lymphoma or grade 3b follicular lymphoma. Monoclonal antibodies, such as pembrolizumab and rituximab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab together with combination chemotherapy may be with a better treatment for diffuse large B-cell lymphoma or follicular lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the toxicity profile of pembrolizumab (MK-3475) when co-administered with full-course RCHOP (rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone) in subjects with previously untreated diffuse large B-cell lymphoma (DLBCL).

SECONDARY OBJECTIVES:

I. To assess clinical outcomes including response rate, event-free survival, and overall survival after MK-3475 + RCHOP induction for subjects with previously untreated DLBCL.

TERTIARY OBJECTIVES:

I. To measure baseline expression of proteins in the programmed death-1 (PD-1) family on tumor cells and coexisting immune infiltrates, using archival tissue when available.

II. To measure peripheral blood T cell subsets before and after treatment using flow cytometry, and to measure baseline vitamin D (25-hydroxy, total).

III. To explore relationships with these parameters and likelihood of response to therapy and outcomes.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and prednisone orally (PO) on days 1-5. Patients also receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 2 of course 1 and on day 1 of subsequent courses. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of the study treatment, patients are followed up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated diffuse large B-cell lymphoma or grade 3B follicular lymphoma (of any stage); subjects must be planned to receive full course (6 cycles) of RCHOP chemoimmunotherapy as per clinical standard of care; patients may have de novo DLBCL, and /or any of the following:

  * Composite lymphomas, which include both diffuse DLBCL and another histology (most commonly follicular lymphoma) in the same lymph node
  * Transformed lymphoma with DLBCL histology, as long as the patient has not received prior therapy for lymphoma
  * Discordant presentations, such as DLBCL in a lymph node and low-grade lymphoma such as follicular lymphoma in the bone marrow
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable nodal disease, including at least 1 disease site measuring 1.5 cm in longest dimension on computed tomography (CT) or fludeoxyglucose (FDG)-positron emission tomography (PET)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale (PS)
* Absolute neutrophil count (ANC) >= 1,500/mcL except in cases of marrow infiltration by lymphoma
* Platelets >= 100,000/mcL except in cases of marrow infiltration by lymphoma
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L except in cases of marrow infiltration by lymphoma
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 ml/min for subject with creatinine levels > 1.5 X institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN or =< 5 X ULN for subjects with liver metastases
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy; as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants; activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy; as long as PT or PTT is within therapeutic range of intended use of anticoagulants, or subject is shown to have an antiphospholipid antibody on workup
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of barrier contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study drug or using an investigation device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* No active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has history of non-infectious pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring intravenous antibiotic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-programmed cell death ligand 1 (PD-L1), anti-programmed cell death ligand 2 (PD-L2), anti-tumor necrosis factor receptor superfamily, member 9 (CD137), or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus surface protein antigen [HBsAg] reactive or hepatitis B virus [HBV] deoxyribonucleic acid [DNA] detectable) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Smith, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab, Combination Chemotherapy): Patients will receive pembrolizumab IV over 30 minutes on day 1 and prednisone PO on days 1-5. Patients also receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 2 of course 1 and on day 1 of subsequent courses. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Cyclophosphamide: Given IV
  Doxorubicin Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Prednisone: Given PO
  Rituximab: Given IV
  Vincristine Sulfate: Given IV
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Combination Chemotherapy)
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Combination Chemotherapy)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 60 [22 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4
  Race: White | 26
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Grade 3 or Higher Toxicity Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The Primary Outcome measures toxicity, with particular attention to Events of Clinical Interest when adding MK-3475 to standard RCHOP therapy. The sample size of 30 patients will permit the estimation of a 40% incidence of grade 3-5 clinically relevant toxicity.
Time Frame: Up to 90 days after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Combination Chemotherapy)
Number analyzed (Participants) | 30
Participants | 13

2. Secondary Outcome: Treatment-related Mortality
Time Frame: Up to 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Event-free Survival
Description: Statistical analysis will entail descriptive statistics, and survival analysis including Kaplan-Meier estimates, log-rank testing of univariate prognostic factors, Cox proportional hazards analysis, as well as T-testing and regression analysis for comparing continuous variables in correlative study data.
Time Frame: Time from diagnosis until relapse or progression, non-protocol re-treatment of lymphoma, or death as a result of any cause, assessed up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Description: as for outcome 3
Time Frame: Date of diagnosis to death from any cause, assessed up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Response Rate Measured by Tumor Imaging
Description: Tumor imaging at baseline and 4-6 weeks, +/-7 days, after 6 courses of induction therapy with MK-3475 + RCHOP to determine remission status. Response will be measured according to 2014 Criteria ("The Lugano Classification").
Time Frame: Up to 6 weeks after course 6
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in T-cell Subsets
Description: Tissue-based assays for tumor and immune infiltrate will be conducted centrally when archival tissue is available. These analyses will seek to identify alterations in T-cell subsets for comparison with historical studies, and exploration of association with treatment outcomes achieved with study therapy.
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the consent form was signed though 90 days following cessation of MK-3475 treatment.
Arm/Group | Treatment (Pembrolizumab, Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Combination Chemotherapy) (N=30)
Upper GI Bleed (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Fever (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection-RSV (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rigors (General disorders) | 1 (1)
Worsening Systolic Function (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Combination Chemotherapy) (N=30)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Syncope (Nervous system disorders) | 3 (3)
Infection (Infections and infestations) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Pulmonary Embolis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Fatigue (General disorders) | 19 (22)
Sensory Neuropathy (Nervous system disorders) | 17 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Constipation (Gastrointestinal disorders) | 12 (12)
Nausea (Gastrointestinal disorders) | 13 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (14)
Dysgeusia (Nervous system disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Abdominal Pain (Gastrointestinal disorders) | 9 (10)
Headache (Nervous system disorders) | 9 (10)
Rash (Skin and subcutaneous tissue disorders) | 9 (9)
Fever (General disorders) | 7 (10)
Dizziness (Nervous system disorders) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Mucositis (Gastrointestinal disorders) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 5 (5)
Dry Mouth (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/65/NCT02541565/Prot_SAP_000.pdf